CLINICAL TRIAL: NCT05761639
Title: Physical Exercise and Telephone Follow-up Mediated by Cardiac Telerehabilitation in Patients With Heart Failure
Brief Title: Physical Exercise and Telephone Follow-up Mediated by Telerehabilitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica de Occidente S.A (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0003
Record Dates: First submitted 2023-02-06; First posted 2023-03-09 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Failure
Keywords: Rehabilitation; telerehabilitation
MeSH Terms: conditions — Heart Failure | interventions — Educational Status; Telerehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telerehabilitation, Education and Telephone Monitoring. (Experimental): The effects of a physical exercise program and educational component with telephone follow-up mediated by cardiac telerehabilitation in patients with heart failure on functional capacity, depression and health-related quality of life will be determined.
  Each participant will be given a polar FT4 brand frequency monitor to record their HR, an OMRON brand digital blood pressure monitor to monitor blood pressure and the conventional Borg scale will be used for perception of exertion during exercise.
  Interventions: Behavioral: Education; Other: telerehabilitation; Behavioral: follow-up
- conventional rehabilitation and Education (Experimental): The effects of a physical exercise program and a conventional educational component in patients with heart failure on functional capacity, depression and health-related quality of life will be determined. The development of this program will be carried out in person guided by a physiotherapist specializing in cardiac and pulmonary rehabilitation.
  Interventions: Other: conventional rehabilitation; Behavioral: Education
- Telerehabilitation and Education (Experimental): To determine the effects of a physical exercise program and a conventional educational component mediated by cardiac telerehabilitation in patients with heart failure on functional capacity, depression, and health-related quality of life
  Each participant will be given a polar FT4 brand frequency monitor to record their HR, an OMRON brand digital blood pressure monitor to monitor blood pressure and the conventional Borg scale will be used for perception of exertion during exercise.
  Interventions: Behavioral: Education; Other: telerehabilitation

INTERVENTIONS:
Other: conventional rehabilitation — The program will be attended in person in the clinic's cardiac rehabilitation program and consists of physical exercise supervised by a physiotherapist specializing in cardiac and pulmonary rehabilitation, for 60 minutes, 3 times a week for a period of 12 weeks, structured by warming up. , muscle strengthening of lower and upper limbs, continuous aerobic training and return to calm.
  Arms: conventional rehabilitation and Education
Behavioral: Education — 1 time a week 30 minutes for each patient individually and in a group with topics: knowledge of the disease, use of medications, warning signs, anxiety management, relaxation techniques, exercises at home, sexual relations and adequate nutrition
Other: telerehabilitation — The program will be assisted by virtual technology and consists of physical exercise at home (for 60 minutes, 3 times a week for a period of 12 weeks, structured by warming up, muscle strengthening of lower and upper limbs, continuous aerobic training and cool down ) supervised by a physiotherapist specializing in cardiac and pulmonary rehabilitation through the "Google Meet" platform
  Arms: Telerehabilitation and Education; Telerehabilitation, Education and Telephone Monitoring.
Behavioral: follow-up — Telephone calls will be made 3 times a week as a follow-up method to obtain information from each person about their heart rate and perception of effort in relation to the activities carried out where they are encouraged to exercise at home on days without intervention.
  Arms: Telerehabilitation, Education and Telephone Monitoring.

SUMMARY:
Cardiovascular diseases are the leading cause of death and disability globally, accounting for approximately 31% (17.9 million) of all deaths each year. The COVID-19 pandemic has led to the total suspension of most cardiac rehabilitation programs at the highest peaks of the spread, forcing people not to leave home, enhancing metabolic conditions and generating further complications due to sedentary lifestyle. Physical exercise is an essential component in the rehabilitation of patients with heart failure disease, evidencing improvements in quality of life, functional capacity, in addition to reducing the mortality rate, number of rehospitalizations, and levels of depression. It is necessary to carry out interventions adapted to the needs of patients who have difficulties traveling to health centers, however, some authors report that remotely oriented exercise could present results similar to those of traditional rehabilitation in a center or Therefore, promoting a cardiac telerehabilitation program together with telephone educational follow-up could cause greater improvements compared to other cardiac rehabilitation and telerehabilitation programs.

Objective: To determine the effects of a physical exercise program and telephone educational follow-up mediated by cardiac telerehabilitation in patients with heart failure on functional capacity, depression, and health-related quality of life.

DETAILED DESCRIPTION:
A randomized controlled clinical trial type study will be carried out, in a period of 6 months between the year 2022, in patients with a diagnosis of heart failure who enter a cardiac rehabilitation program in the city of Santiago de Cali, Colombia, linking to the research after the consultation with cardiology in three groups: physical exercise program and conventional educational component with telephone follow-up (Intervention), physical exercise program and conventional educational component mediated by cardiac telerehabilitation, to which measurements of sociodemographic variables and clinical before-after measurements (physiological, paraclinical, anthropometric) functional capacity, quality of life and state of depression.

ELIGIBILITY:
Inclusion Criteria:

* patients previously diagnosed by a Cardiology Specialist with heart failure.
* Patients who present an indication to exercise.
* Patients who have digital equipment such as a computer, tablet or cell phone with access to virtual platforms to carry out exercise sessions mediated by technology.
* Participants who accept and sign the informed consent.

Exclusion Criteria:

* Patients with respiratory comorbidity or who present some limitation to perform active and resisted movements (recent fractures, recent hemodynamic alterations, coronary disease event after the diagnosis of cardiovascular disease, infectious diseases and neuromuscular limitation).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Adherence to exercise | measured 6 months after the intervention
  Practicing physical activity as a principle of self-determination and converting it into a healthy lifestyle or habit and aerobic capacity will be measured by completing 85% of sessions (21 sessions) of cardiac rehabilitation, including education and telephone follow-up.
health-related quality of life | measured 6 months after the intervention
  A generic concept that reflects the concern for the modification and improvement of the attributes of life, for example, the physical, political, moral, social environment, as well as health and disease.
  It is applied with the Saint George's Questionnaire (SGRQ), this scale goes from 0 to 100 points, high scores indicate that the patient is unwell and low scores the patient is better and a decrease of 4 points after an intervention is considered clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Jhonatan Betancourt Peña, PT, Principal Investigator — Institucion Universitaria Escuela Nacional del Deporte - Universidad de Vigo
Locations (1):
- Programa de Rehabilitacion, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Enfermedades Cardiovasculares. Prevención y control de las enfermedades no transmisibles [Internet]. OMS. 2016 [citado 19 octubre 2021]. Disponible en: https://www.paho.org/es/temas/enfermedades-cardiovasculares. Organización Mundial de la Salud. Estrategia mundial para la prevención y el control de las enfermedades no transmisibles. 2000
- [Background] Piotrowicz E, Pencina MJ, Opolski G, Zareba W, Banach M, Kowalik I, Orzechowski P, Szalewska D, Pluta S, Glowczynska R, Irzmanski R, Oreziak A, Kalarus Z, Lewicka E, Cacko A, Mierzynska A, Piotrowicz R. Effects of a 9-Week Hybrid Comprehensive Telerehabilitation Program on Long-term Outcomes in Patients With Heart Failure: The Telerehabilitation in Heart Failure Patients (TELEREH-HF) Randomized Clinical Trial. JAMA Cardiol. 2020 Mar 1;5(3):300-308. doi: 10.1001/jamacardio.2019.5006. PMID 31734701
- [Background] Tersalvi G, Winterton D, Cioffi GM, et al. Telemedicina en insuficiencia cardíaca durante COVID-19: un paso hacia el futuro. Delantero Cardiovasc Med . 2020;7:612818. Publicado el 9 de diciembre de 2020. doi:10.3389/fcvm.2020.612818
- [Background] Piotrowicz E, Stepnowska M, Leszczynska-Iwanicka K, Piotrowska D, Kowalska M, Tylka J, Piotrowski W, Piotrowicz R. Quality of life in heart failure patients undergoing home-based telerehabilitation versus outpatient rehabilitation--a randomized controlled study. Eur J Cardiovasc Nurs. 2015 Jun;14(3):256-63. doi: 10.1177/1474515114537023. Epub 2014 May 21. PMID 24849304
- [Background] Brouwers RWM, van Exel HJ, van Hal JMC, Jorstad HT, de Kluiver EP, Kraaijenhagen RA, Kuijpers PMJC, van der Linde MR, Spee RF, Sunamura M, Uszko-Lencer NHMK, Vromen T, Wittekoek ME, Kemps HMC; Committee for Cardiovascular Prevention and Cardiac Rehabilitation of the Netherlands Society of Cardiology. Cardiac telerehabilitation as an alternative to centre-based cardiac rehabilitation. Neth Heart J. 2020 Sep;28(9):443-451. doi: 10.1007/s12471-020-01432-y. PMID 32495296
- [Background] Frederix I, Hansen D, Coninx K, et al. Telerehabilitación III: un ensayo multicéntrico, aleatorizado y controlado que investiga la eficacia a largo plazo de un programa integral de telerehabilitación cardíaca: justificación y diseño del estudio. Trastorno cardiovascular BMC . 2015;15:29. Publicado el 7 de mayo de 2015. doi:10.1186/s12872-015-0021-5
- [Background] Hwang R, Bruning J, Morris NR, Mandrusiak A, Russell T. Home-based telerehabilitation is not inferior to a centre-based program in patients with chronic heart failure: a randomised trial. J Physiother. 2017 Apr;63(2):101-107. doi: 10.1016/j.jphys.2017.02.017. Epub 2017 Mar 14. PMID 28336297
- [Background] Bernocchi P, Vitacca M, La Rovere MT, Volterrani M, Galli T, Baratti D, Paneroni M, Campolongo G, Sposato B, Scalvini S. Home-based telerehabilitation in older patients with chronic obstructive pulmonary disease and heart failure: a randomised controlled trial. Age Ageing. 2018 Jan 1;47(1):82-88. doi: 10.1093/ageing/afx146. PMID 28985325
- [Background] Peng X, Su Y, Hu Z, Sun X, Li X, Dolansky MA, Qu M, Hu X. Home-based telehealth exercise training program in Chinese patients with heart failure: A randomized controlled trial. Medicine (Baltimore). 2018 Aug;97(35):e12069. doi: 10.1097/MD.0000000000012069. PMID 30170422
- [Background] Tam CF, Cheung KS, Lam S, Wong A, Yung A, Sze M, Lam YM, Chan C, Tsang TC, Tsui M, Tse HF, Siu CW. Impact of Coronavirus Disease 2019 (COVID-19) Outbreak on ST-Segment-Elevation Myocardial Infarction Care in Hong Kong, China. Circ Cardiovasc Qual Outcomes. 2020 Apr;13(4):e006631. doi: 10.1161/CIRCOUTCOMES.120.006631. Epub 2020 Mar 17. No abstract available. PMID 32182131
- [Background] Tersalvi G, Winterton D, Cioffi GM, Ghidini S, Roberto M, Biasco L, Pedrazzini G, Dauw J, Ameri P, Vicenzi M. Telemedicine in Heart Failure During COVID-19: A Step Into the Future. Front Cardiovasc Med. 2020 Dec 9;7:612818. doi: 10.3389/fcvm.2020.612818. eCollection 2020. PMID 33363223
- [Background] Kikuchi A, Taniguchi T, Nakamoto K, Sera F, Ohtani T, Yamada T, Sakata Y. Feasibility of home-based cardiac rehabilitation using an integrated telerehabilitation platform in elderly patients with heart failure: A pilot study. J Cardiol. 2021 Jul;78(1):66-71. doi: 10.1016/j.jjcc.2021.01.010. Epub 2021 Feb 10. PMID 33579602
- [Background] Osorio MAM. Del Modelo Biomédico al Modelo Biopsicosocial: El desafío pendiente para la fisioterapia en el dolor músculoesquelético crónico. Revista Facultad de Ciencias de la Salud UDES. 2016;3(2):97-101.
- [Derived] Betancourt-Pena J, Portela-Pino I, Martinez-Patino MJ. Study protocol for a controlled clinical trial on cardiac telerehabilitation and educational follow-up in patients with heart failure. PLoS One. 2025 Jul 10;20(7):e0327366. doi: 10.1371/journal.pone.0327366. eCollection 2025. PMID 40638607